CLINICAL TRIAL: NCT03450317
Title: The Influence of Aspirin on Human Gut Microbiota Composition and Metabolome: Contributing to the Therapeutic Effects of the Drug
Brief Title: Influence of Aspirin on Human Gut Microbiota Composition and Metabolome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Francis KL Chan, Prof. Francis Chan, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ASP MIC study
Record Dates: First submitted 2018-02-22; First posted 2018-03-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Aspirin; Microbiota
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin (Experimental): Aspirin 80mg once daily
  Interventions: Drug: Aspirin 80mg
- Non-treatment group (No Intervention): No intervention

INTERVENTIONS:
Drug: Aspirin 80mg — No treatment
  Other Names: Non-treatment
  Arms: Aspirin

SUMMARY:
Colorectal cancer (CRC) is the third most common cancer type in males and the second in females, accounting for about 693,900 deaths worldwide per year. Although the annual CRC mortality rate is still very high, it demonstrated a decline by 47% among men and 44% among women from 1990 to 2015. This decreasing trend may be attributed to improved screening, early detection as well as combined CRC treatment. In fact, the mortality rate is expected to reduce further by long-term use of chemopreventive agents that can prevent the development of neoplasms in the large bowel. Several decades of research both in clinic and laboratory has identified aspirin as an effective synthetic CRC chemoprevention drug.

It is commonly accepted that aspirin exerts its chemopreventive effects by inhibiting catalytic enzymes cyclooxygenase (COX) -1 and COX-2 involved in prostaglandin synthesis. But the mechanism of its chemopreventive effect on CRC is not clearly understood. Other than CRC, aspirin also showed its potential inhibitory effects on some other types of solid cancer, such as pancreatic, lung, breast and prostate cancers. However, its effects on extragastrointestinal cancer types are still elusive due to lack of reliable supporting evidence from randomized clinical trials. Based on current knowledge, it is unclear why aspirin appears to inhibit CRC more than other cancers. This might be associated with the unique microenvironment comprising trillions of microbes in which CRC resides.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common cancer type in males and the second in females, accounting for about 693,900 deaths worldwide per year.

It is commonly accepted that aspirin exerts its chemopreventive effects by inhibiting catalytic enzymes cyclooxygenase (COX) -1 and COX-2 involved in prostaglandin synthesis.This hypothetic mechanism is supported by clinical data from two large cohorts that found that the regular use of aspirin reduced the risk of CRC with high expression of COX-2 but not with low or no expression of COX-2.

Based on current knowledge, it is unclear why aspirin appears to inhibit CRC more than other cancers. This might be associated with the unique microenvironment comprising trillions of microbes in which CRC resides. Therefore, the investigator hypothesizes that there is a link between the chemopreventive mechanism of aspirin, gut microbiota as well as the metabolome.

During the past decade, evidence has accumulated that microbiota in the host is highly sensitive to the gut microenvironment since its composition and activity can be rapidly and reproducibly changed by diet or nutrients. As such, an acidic drug like aspirin may be able to alter the gut microbiota composition. It is thus conceivable that the CRC preventive action of aspirin may be through the alteration of host gut microbes.

ELIGIBILITY:
Inclusion Criteria:

* NSAID naïve during the last month;
* absence of drugs, nutrient supplements, probiotics, prebiotics and synbiotics that might interfere with microbial homeostasis for all participants;
* no past history of gastrointestinal bleeding or ulcers;
* absence of historical aspirin-induced side effects;
* voluntary and willing to cooperate during treatment; and
* consent with treatment and sample collection schedule

Exclusion Criteria:

* unfit symptoms, such as epigastric pain, acid reflux, eructation and dyspepsia;
* diagnosis of any disease during the past 3 months;
* diarrhea within the previous 7 days;
* history of alcohol abuse, defined as >80 g/d in men and >40 g/d in women;
* pregnancy; and
* mental illness rendering the participants unable to understand the nature, scope, and possible consequences of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
gut microbiota in stool | 1 year
  To capture the fingerprint of gut microbiota in stool before and after oral administration of aspirin
metabolome in biological specimens | 1 year
  To capture the metabolome in biological specimens before and after oral administration of aspirin

SECONDARY OUTCOMES:
gut microbial composition | 1 year
  To profile the alteration of gut microbial composition by aspirin
metabolomic components | 1 year
  To profile the alteration of the metabolomic components by aspirin

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong